CLINICAL TRIAL: NCT03497884
Title: Individualized Precise Localization of rTMS on Primary Motor Area and Its Effects on Basal Ganglia
Brief Title: Individualized Precise Localization of rTMS on Primary Motor Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Yu-Feng ZANG, Professor, Hangzhou Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HZNU_initiative_movement_rTMS
Record Dates: First submitted 2017-09-07; First posted 2018-04-13 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease
Keywords: fMRI; rTMS; functional connectivity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real rTMS (low frequency) (Experimental): Real rTMS (low frequency) is 1Hz.
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator): Sham rTMS session includes low frequency and high frequency stimulations.
  Interventions: Device: rTMS
- Real rTMS (high frequency) (Experimental): Real rTMS (high frequency) is 10Hz.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — For the l-Hz sessions (low frequency), stimulation is delivered at 100% of the subject's resting motor threshold at 1 Hz continuously over 30 min for a total of 1,800 pluses. The 10-Hz stimulation (high frequency) is delivered at 100% of the subject's resting motor threshold via 60 trains of 3-s 10-Hz rTMS (30 pulses per train).

SUMMARY:
Parkinson's disease (PD) patients have some problem with self-initiated movement task. Compared with health controls, task meta-analysis found that PD patients showed abnormal activation in pre-supplementary motor area (pre-SMA) and putamen. And the functional connectivity has already been reported between pre-SMA and putamen in 2013. Repetitive Transcranial Magnetic Stimulation (rTMS) is a sage and painless technique to activate cortical areas. The deep brain structure can be activated via stimulating superficial cortex by rTMS. For investigating the mechanism of self-initiated movement, this project is using functional magnetic resonance imaging (fMRI) to individualize the precise localization in motor area and combining rTMS to activate putamen.

DETAILED DESCRIPTION:
Healthy subject is recruiting in this project. High and low frequency rTMS will be performed, respectively. For the l-Hz sessions (low frequency), stimulation is delivered at 100% of the subject's resting motor threshold at 1 Hz continuously over 30 min for a total of 1,800 pluses. The 10-Hz stimulation is delivered at 100% of the subject's resting motor threshold via 60 trains of 3-s 10-Hz rTMS (30 pulses per train).

ELIGIBILITY:
Inclusion Criteria:

* There are activation in motor area during the task fMRI
* The head motion less than 2 mm in translation or 2 degrees in rotation in any direction during the resting-state fMRI

Exclusion Criteria:

* Without any neuropsychiatric conditions
* No head injury or history of epilepsy
* Not on any medications

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
degree of enhanced neuro-activity associated with frequency-specific treatment | through study completion, an average of 1 year
  functional connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Feng Zang, M.D., Principal Investigator — Hangzhou Normal University
Locations (2):
- China (2):
  - Hangzhou Normal University,Center for Cognition and Brain Disorder, Hangzhou, Zhejiang
  - Hangzhou Normal University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang JX, Rogers LM, Gross EZ, Ryals AJ, Dokucu ME, Brandstatt KL, Hermiller MS, Voss JL. Targeted enhancement of cortical-hippocampal brain networks and associative memory. Science. 2014 Aug 29;345(6200):1054-7. doi: 10.1126/science.1252900. PMID 25170153
- [Result] Eldaief MC, Halko MA, Buckner RL, Pascual-Leone A. Transcranial magnetic stimulation modulates the brain's intrinsic activity in a frequency-dependent manner. Proc Natl Acad Sci U S A. 2011 Dec 27;108(52):21229-34. doi: 10.1073/pnas.1113103109. Epub 2011 Dec 12. PMID 22160708